CLINICAL TRIAL: NCT04688112
Title: A Validation Study Comparing the Heart Rate, Respiratory Rate, Heart Rate Variability and Blood Pressure Obtained by Video Selfie Using the DocMe® Technology With Those Obtained by Direct Measurement in Healthy People
Brief Title: Validation Study of Selfie Technology for Assessment of Vital Signs
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: DocMe Technologies Ltd (Industry)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PRFX-2020-01-DocMe
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Photoplethysmography; Video Selfie; Vital Signs; Blood Pressure; Smartphone; DocMe; Heart Rate; Respiratory Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to compare accuracy of DocMe, a video technology developed by DocMe Health Technologies, with previously validated medical devices used for measurements of heart rate, heart rate variability, respiratory rate and blood pressure in adults.

DETAILED DESCRIPTION:
Photoplethysmography (PPG) makes uses of low-intensity infrared (IR) light. When light travels through biological tissues, it is absorbed by bones, skin pigments and both venous and arterial blood. However, as light is more strongly absorbed by blood than the surrounding tissues, the changes in blood flow can be detected by PPG sensors as changes in the intensity of light.

The signal from PPG is proportional to the quantity of blood flowing through the blood vessels and even small changes in blood volume can be detected using this method. Analysis of the waveform can provide information on a range of physiological measurements affecting the cardiovascular and respiratory systems. PPG is widely used in medicine in the form of pulse oximeters using sensors applied to peripheral digits.

Recently, it has been shown that PPG data can be obtained using images acquired from videos taken using the camera on smartphones and there is now a significant and growing body of published literature to support this.

DocMe Health Technologies has developed a system of obtaining these data using a 15 second video selfie.

At this time, the technology has been shown to be reasonably accurate when compared to home devices in healthy subjects. However, to make the technology more widely useful, the results obtained by video selfies need to be formally validated.

The aim of the study therefore is to compare measurements obtained from video selfies with measurements taken using already validated machines in the same patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 - 90 years old).
* Participants must be willing and able to give informed consent for participation in the study, and considered fit for the study by the nurse.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will seek to adhere to ISO (81060-2:2018)guidelines and AHA BP consensus standards.
  * at least 5% population reference range systolic BP <100mmHg
  * at least 5% population reference range systolic BP >160mmHg
  * at least 20% population reference range systolic BP >140mmHg
  * at least 5% population reference range diastolic BP <60mmHg
  * at least 5% population reference range diastolic BP >100mmHg
  * at least 20% population reference range diastolic BP >80mmHg
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | Baseline
  Heart Rate (beats/minute) assessed 3 times at 10 minute intervals on one occasion
Respiratory Rate | Baseline
  Respiratory Rate in respirations/min assessed visually or oximeter if it has the capability assessed 3 times at 10 minute intervals on one occasion
Heart Rate Variability | Baseline
  HRV (ms) assessed 3 times at 10 minute intervals on one occasion
Blood Pressure | Baseline
  Systolic and Diastolic Blood Pressure assessed 3 times at 10 minute intervals on one occasion

CONTACTS AND LOCATIONS:
Overall Officials: Alex T Novak, MRCGP FRCEM, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barszczyk A, Lee K. Measuring Blood Pressure: from Cuff to Smartphone. Curr Hypertens Rep. 2019 Oct 10;21(11):84. doi: 10.1007/s11906-019-0990-3. PMID 31599362
- [Background] Luo H, Yang D, Barszczyk A, Vempala N, Wei J, Wu SJ, Zheng PP, Fu G, Lee K, Feng ZP. Smartphone-Based Blood Pressure Measurement Using Transdermal Optical Imaging Technology. Circ Cardiovasc Imaging. 2019 Aug;12(8):e008857. doi: 10.1161/CIRCIMAGING.119.008857. Epub 2019 Aug 6. PMID 31382766
- [Background] Chowdhury MH, Shuzan MNI, Chowdhury MEH, Mahbub ZB, Uddin MM, Khandakar A, Reaz MBI. Estimating Blood Pressure from the Photoplethysmogram Signal and Demographic Features Using Machine Learning Techniques. Sensors (Basel). 2020 Jun 1;20(11):3127. doi: 10.3390/s20113127. PMID 32492902
- [Background] Humphreys K, Ward T, Markham C. Noncontact simultaneous dual wavelength photoplethysmography: a further step toward noncontact pulse oximetry. Rev Sci Instrum. 2007 Apr;78(4):044304. doi: 10.1063/1.2724789. PMID 17477684
- [Background] Kong L, Zhao Y, Dong L, Jian Y, Jin X, Li B, Feng Y, Liu M, Liu X, Wu H. Non-contact detection of oxygen saturation based on visible light imaging device using ambient light. Opt Express. 2013 Jul 29;21(15):17464-71. doi: 10.1364/OE.21.017464. PMID 23938616